CLINICAL TRIAL: NCT00086710
Title: An Open-label, Randomized, Cross-over Study in HIV-Positive Subjects to Determine and Compare the Single-dose Pharmacokinetics of Enfuvirtide after a Single 90 mg SC Administration
Brief Title: Study of Enfuvirtide in HIV-Positive Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trimeris (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: T20-405
Record Dates: First submitted 2004-07-08; First posted 2004-07-13 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-04

CONDITIONS: HIV Infections; AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Enfuvirtide

INTERVENTIONS:
Drug: Fuzeon

SUMMARY:
A total of 26 patients will be admitted to the clinic where they will be dosed with each injection device. There will be a 7-day washout between doses and a 7-10 day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26

CONTACTS AND LOCATIONS:
Locations (1):
- SFBC, Miami, Florida, United States